CLINICAL TRIAL: NCT02000596
Title: 1303GCC: Phase II Study of Trastuzumab and Pertuzumab Alone and in Combination With Hormonal Therapy or Chemotherapy in Women Aged 60 and Over With HER2/Neu Overexpressed Locally Advanced and/or Metastatic Breast Carcinoma
Brief Title: 1303GCC: Trastuzmab & Pertuzumab With Hormonal Therapy or Chemotherapy in Women Aged 60 and Over.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding withdrawn by sponsor
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00054959; 1303GCC; GCC1303 (Other: University of Maryland Greenebaum Cancer Center)
Record Dates: First submitted 2013-11-21; First posted 2013-12-04 (Estimated); Results first posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2 overexpressed; Metastatic Breast Cancer; Elderly
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; Anastrozole; Fulvestrant; Drug Therapy; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1: T+P (Experimental): Trastuzumab plus Pertuzumab as first line treatment for HER2 overexpressed Metastatic Breast Cancer (without hormonal therapy or chemotherapy)
  Interventions: Drug: Trastuzumab plus Pertuzumab
- Cohort 2 - Arm A (Experimental): Hormonal Therapy with Anastrozole and Fulvestrant in addition Trastuzumab plus Pertuzumab for women who progressed on T+P alone, and who are ER/PR +
  Interventions: Drug: Trastuzumab plus Pertuzumab; Drug: Hormonal Therapy with Anastrozole and Fulvestrant
- Cohort 2 - Arm B (Experimental): Chemotherapy with Eribulin in addition to Trastuzumab plus Pertuzumab for women who progressed on T+P alone and who are ER/PR -
  Interventions: Drug: Trastuzumab plus Pertuzumab; Drug: Chemotherapy with Eribulin

INTERVENTIONS:
Drug: Trastuzumab plus Pertuzumab
Drug: Hormonal Therapy with Anastrozole and Fulvestrant — Anastrozole 1mg by mouth daily FULVESTRANT 500mg i.m. D1, D15, D28 then every 28-30 days
  Other Names: Anastrozole (Arimidex); Fulvestrant (Faslodex)
  Arms: Cohort 2 - Arm A
Drug: Chemotherapy with Eribulin
  Arms: Cohort 2 - Arm B

SUMMARY:
This is a phase II study that combines Trastuzumab with Pertuzumab to see how it works in women age greater than 60 who have been diagnosed with HER2/neu overexpressed locally advanced and/or metastatic breast carcinoma.

DETAILED DESCRIPTION:
Currently available standard therapies for HER2 overexpressed metastatic breast cancers (MBC) include treatments with chemotherapy or hormonal therapy, alone or in combination with medications that target HER2 gene, such as Trastuzumab or Pertuzumab. This study will examine the effect of treating HER2 overexpressed MBC with the combination of Trastuzumab plus Pertuzumab, without hormonal or chemotherapy, as a first line treatment. If patients progress on this treatment, they will receive hormonal or chemotherapy in addition to the Trastuzumab plus Pertuzumab treatment. The objective is to see how the overall response rate for this treatment compares to other first line treatments in the same patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥60 Years of Age.
2. Histologically confirmed, locally advanced (T4 primary tumor and stage IIIB or IIIC disease) or metastatic breast cancer that progressed after treatment with standard treatment regimens in the adjuvant or neoadjuvant setting.
3. Prior treatment with trastuzumab and/or lapatinib in the neo-adjuvant or adjuvant setting is allowed but not required. Lapatininb has to be discontinued > 21 days before the initiation of the T+P study treatments.
4. Up to 3 prior chemo regimens for treatment of metastatic disease are allowed as long as the study subject is acceptable for study treatment with chemo required on this study in cohort 2 at progression on T+P.
5. Patients may have had prior hormonal therapy with any hormonal agents as per section 3.1.5 of this protocol.
6. Zometa or denosumab can be continued as per standard of care as long as started before the study treatment is started.
7. HER2 positive breast cancer, as defined in Section 3.3 of this protocol
8. Must have measurable or evaluable disease according to RECIST 1.1 criteria.
9. Lab values obtained ≤7 days prior to registration as indicated in 3.1.9 of this protocol.
10. ECOG Performance Status (PS) of 0, 1 or 2.
11. LVEF at least 50% as determined by MUGA or ECHO.
12. Life expectancy >3 months.
13. Written informed consent.
14. Willingness to return to study site for treatment and follow-up.
15. Normal QTc interval defined on EKG as QTc ≤ 440 msec.
16. Postmenopausal women defined in section 3.1.16 of this protocol.

Exclusion Criteria:

1. Stage III or IV cancer, other than breast cancer, in ≤5 years prior to registration.
2. Actively being treated for other malignancy.
3. New York Heart Association Class III or IV cardiovascular disease.
4. History of coronary heart failure (CHF)
5. Current use of drugs known to prolong the QTc interval including Class Ia and III antiarrhythmics or history of congenital long QTc syndrome.
6. Evidence of active brain metastasis including leptomeningeal involvement.
7. Major surgery, chemotherapy, hormonal or immunologic therapy ≤3 weeks prior to registration.
8. Radiotherapy ≤3 weeks prior to registration, except if to a non-target lesion only.
9. Prior treatment with Pertuzumab, Eribulin, Fulvestrant or Anastrozole.
10. Uncontrolled illness.
11. Co-morbid systemic illnesses or other severe concurrent disease. See section 3.2.11.
12. Currently receiving treatment in a different clinical study in which investigational procedures are performed or investigational therapies are administered.
13. Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be HIV positive.
14. International normalized ratio (INR), activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) >1.5 × ULN (unless on anticoagulation medication)
15. Receipt of intravenous (IV) antibiotics for infection within 7 days prior to enrollment into the study.
16. Current chronic daily treatment with corticosteroids. See section 3.2.16 of this protocol.
17. Known hypersensitivity to any of the study treatments or to excipients of recombinant human or humanized antibodies.
18. History of receiving any investigational treatment within 28 days prior to enrollment into the study.
19. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Tkaczuk, MD, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (1):
- University of Maryland Marlene & Stewart Greenebaum Cancer Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: T+P: Trastuzumab plus Pertuzumab as first line treatment for HER2 overexpressed Metastatic Breast Cancer (without hormonal therapy or chemotherapy)
  Trastuzumab plus Pertuzumab
- Cohort 2 - Arm A: Hormonal Therapy with Anastrozole and Fulvestrant in addition Trastuzumab plus Pertuzumab for women who progressed on T+P alone, and who are ER/PR +
  Trastuzumab plus Pertuzumab
  Hormonal Therapy with Anastrozole and Fulvestrant: Anastrozole 1mg by mouth daily FULVESTRANT 500mg i.m. D1, D15, D28 then every 28-30 days
- Cohort 2 - Arm B: Chemotherapy with Eribulin in addition to Trastuzumab plus Pertuzumab for women who progressed on T+P alone and who are ER/PR -
  Trastuzumab plus Pertuzumab
  Chemotherapy with Eribulin
Period: Cohort 1
Arm/Group | Cohort 1: T+P | Cohort 2 - Arm A | Cohort 2 - Arm B
Started | 2 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Cohort 2
Arm/Group | Cohort 1: T+P | Cohort 2 - Arm A | Cohort 2 - Arm B
Started | 0 | 0 | 2
Completed | 0 | 0 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants started in "Cohort 1: T+P" Arm/Group and continued in "Cohort 2 Arm B" due to progressive disease
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: T+P | Cohort 2 - Arm A | Cohort 2 - Arm B | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0 | 0
  Between 18 and 65 years | 2 |  | 0 | 2
  >=65 years | 0 |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 0 | 2
  Male | 0 |  | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/ Non-Hispanic | 2 |  | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) in Patients
Description: Defined as the total of complete response (CR) defined as a disappearance of all target lesions, partial response (PR) defined as >= 30% decrease in the sum of the longest diameter of target lesions, and stable disease (SD) >= 27 weeks among the total number of participants as defined by the Response Evaluation in Solid Tumors (RECIST) 1.1 response criteria.
Time Frame: Participants were staged every two cycles for the duration of the study participation ( CR+PR+SD=ORR), up to 11 months
Population: Participants started in "Cohort 1: T+P" Arm/Group and continued in "Cohort 2 Arm B" due to progressive disease
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: T+P | Cohort 2 - Arm A | Cohort 2 - Arm B
Number analyzed (Participants) | 2 | 0 | 2
Participants
  Complete Response (CR) | 0 |  | 0
  Partial Response (PR) | 1 |  | 0
  Stable Disease (SD) | 1 |  | 2

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression Free Survival in treatment cohorts 1 and 2 as well as arms A and B from the time on study until progression of disease or death
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 11 months
Population: No participants were enrolled in Cohort 2- Arm A
Measure: Number; unit: weeks
Arm/Group | Cohort 1: T+P | Cohort 2 - Arm A | Cohort 2 - Arm B
Number analyzed (Participants) | 2 | 0 | 2
weeks
  Subject 1 | 6 |  | 12
  Subject 2 | 24 |  | 24

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) in treatment cohorts 1 and 2 as well as arms A and B from the time on study until death
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed through study completion, an average of 2 years.
Population: Participants started in "Cohort 1: T+P" Arm/Group and continued in "Cohort 2 Arm B" due to progressive disease. The analysis below reflects Cohort 2 only
Measure: Number; unit: Months
Arm/Group | Cohort 1: T+P | Cohort 2 - Arm A | Cohort 2 - Arm B
Number analyzed (Participants) | 0 | 0 | 2
Months
  Subject 1 |  |  | 25
  Subject 2 |  |  | 14

4. Secondary Outcome: Number of Participants With Treatment Related Adverse Events as Assessed by CTCAE v4.0
Description: the safety and tolerability of Trastuzumab and Pertuzumab alone and in combination with hormonal therapy or single agent chemotherapy. in HER2+ MBC patients
Time Frame: Participants were followed during the study and for 30 days after completion of the study treatment, up to 12 months
Population: No participants were enrolled in Cohort 2- Arm A
Measure: Number; unit: participants
Arm/Group | Cohort 1: T+P | Cohort 2 - Arm A | Cohort 2 - Arm B
Number analyzed (Participants) | 2 | 0 | 2
participants
  participant 1 | 5 |  | 2
  participant 2 | 5 |  | 8

5. Secondary Outcome: Quality of Life Via Patient-reported Outcomes
Description: quality of life and treatment side effects via patient-reported and investigator reported outcomes
Time Frame: Duration of study, participants were followed every cycle up to 11 months.
Population: Two patients were enrolled, no data was analyzed.
Arm/Group | Cohort 1: T+P | Cohort 2 - Arm A | Cohort 2 - Arm B
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 24 months
Description: There were no participants enrolled in Cohort 2 - Arm A, therefore, the at risk population for all-cause mortality, SAEs, and AEs are zero.
Arm/Group | Cohort 1: T+P | Cohort 2 - Arm A | Cohort 2 - Arm B
All-Cause Mortality (participants affected / at risk) | 2/2 | 0/0 | 2/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: T+P (N=2) | Cohort 2 - Arm A (N=0) | Cohort 2 - Arm B (N=2)
muscle aches or neck aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 1
smell aversion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 1
elevated AST (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) — Grade 1
elevated ALT (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) — Grade 1
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) — Grade 1
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) — Grade 1
Rigors (General disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 2
Paresthia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 1
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 1
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Grade 1
Reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Grade 2
Insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Grade 2
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Grade 2
Taste Changes (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes